CLINICAL TRIAL: NCT02644434
Title: A Randomized Comparison of Conventional Versus Intentional StraTegy in Patients With High Risk PrEdiction of Side Branch OccLusion in Coronary Bifurcation InterVEntion: the CIT-RESOLVE Trial
Brief Title: Conventional Versus Intentional StraTegy in Lesions With High Risk PrEdiction of Side Branch OccLusion in InterVEntion
Acronym: CIT-RESOLVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: China_NCCD
Record Dates: First submitted 2015-12-01; First posted 2015-12-31 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Coronary Bifurcation Intervention; Randomized Clinical Trial
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Strategy (Active Comparator): Patients randomized to the conventional strategy group would undergo either jailed wire technique (diameter of side branch<2.5mm and ≥2.0mm) or provisional two-stent strategy (diameter of side branch≥2.5mm).
  Interventions: Procedure: Conventional Strategy
- Intentional Strategy (Experimental): Patients randomized to the intentional strategy group would undergo either jailed balloon technique (diameter of side branch<2.5mm and ≥2.0mm) or elective two-stent strategy (diameter of side branch≥2.5mm).
  Interventions: Procedure: Intentional strategy

INTERVENTIONS:
Procedure: Conventional Strategy — Jailed wire technique: Both MV and SB are wired. The MV is stented with wire protection in SB. The SB is not further treated unless there is threatened SB closure, severe ostial pinching of SB (>90%), TIMI flow grade decrease in SB, or SB dissection greater than type A. If one of these criteria exists, the SB would be rewired and a kissing balloon inflation is undertaken.
  Provisional two-stent strategy: Lesion preparation and MV stenting are the same as the jailed wire technique. Provisional T stenting of the SB could be undertaken if one of the following criteria exists after SB rewiring and a kissing balloon inflation is undertaken: threatened SB closure, severe ostial pinching of SB (>90%), TIMI flow grade decrease in SB, or SB dissection greater than type A.
  Arms: Conventional Strategy
Procedure: Intentional strategy — Jailed balloon technique: The technique has been detailed in previous studies. A monorail balloon that is angiographically sized to approximate the Side Branch (SB) vessel diameter is advanced into the SB. If there is TIMI flow grade decrease in the SB after MV stenting, the SB balloon is inflated to simulate attempt to reopen the SB. The procedure would be completed with the standard kissing balloon technique no matter there is SB compromise or not.
  Elective two-stent strategy: Patients in this subgroup would undergo crush procedure or any other elective two-stent strategy which stenting SB before MV stenting.
  Arms: Intentional Strategy

SUMMARY:
The purpose of the present study is to investigate if intentional strategy (a more aggressive side branch protection strategy: elective two-stent or jailed balloon technique) is associated with significant reduction of side branch occlusion rate compared to conventional strategy (provisional two-stent strategy or jailed wire technique) in patients at high risk of side branch occlusion (V-RESOLVE score≥12).

DETAILED DESCRIPTION:
1. Statistical Design and Analysis.

   1.1 Analysis Population(s).

   1.1.1 Intent to Treat Population (ITT, primary clinical endpoint only).

   The ITT population set will consist of all subjects who signed the written informed consent and are randomized, regardless which strategy was selected.

   The primary analysis is a superiority ITT analysis of the primary clinical endpoint, being side branch occlusion after main vessel stenting.

   1.1.2 Per Protocol (PP, for clinical endpoints).

   If required, an additional analysis of the Per-Protocol (PP) population will be conducted of the primary and secondary endpoints. The PP population consists of those subjects who correctly received (only) the assigned study stent. Should all subjects correctly receive (only) the assigned study stent(s), no PP analysis will be required for the clinical endpoints.

   1.2 Statistical Methods.

   1.2.1 Statistical Hypothesis for the Primary Endpoint.

   H0: Pt-Pc ≥0;

   H1: Pt-Pc <0;

   where Pt and Pc are the rates of side branch occlusion in the intentional strategy (test) and convention strategy (control) groups, respectively.

   The study is powered at 80% to show differences in the rate of side branch occlusion between intentional strategy group and conventional strategy group. The primary analysis will be performed for the ITT patient population.

   1.2.2 Statistical Test Method for the Primary Endpoint.

   Normal approximation test for the difference between two proportions (pooled proportion) or Fisher's exact test (if applicable) will be used to test the two-sided hypothesis of superiority in proportions. If the P value from the two-sided test is <0.05, the intentional strategy (test) will be concluded to be superior to conventional strategy. This corresponds to the two-sided upper 95% confidence bound on the difference between treatment groups in side branch occlusion (the intentional strategy - conventional strategy) being less than delta.

   1.2.3 Sample Size Parameters for the Primary Endpoint.
   * A 1:1 treatment allocation ratio of intentional strategy group and the conventional strategy group
   * A two-side significance level (alpha) of 0.05
   * 80% power to show differences in the rate of side branch occlusion between intentional strategy group and conventional strategy group
   * The rate of side branch occlusion in intentional strategy group: 4.0%
   * The rate of side branch occlusion in conventional strategy group: 10.0%
   * The primary endpoint would be reached immediately after the main vessel stenting, therefore, the attrition rate is 0%

   The 10% rate of side branch occlusion in conventional strategy group is based on the V-RESOLVE study. It is reasonable to assume that, with an intentional strategy for bifurcation lesions with V-RESOLVE score ≥12 points, the rate of side branch occlusion would decrease to 4% in intentional strategy group. Thus, the present study requires 283 subjects in intentional strategy group and 283 in conventional strategy group, and the total number will be 566.

   1.3 Secondary Endpoint Analysis.

   For all secondary endpoints the results of the intentional strategy and conventional strategy groups will be compared.

   For clinical endpoint the analysis will be performed at each follow-up visit, meaning at 1 Month, 3 Months, 6 Months and 12 Months. The analysis will be performed for the ITT population and, if applicable, the PP population.

   For all secondary endpoints conventional p-values and 95% confidence intervals for the difference in Kaplan-Meier will be calculated.

   Dichotomous variables will be evaluated using Fisher's exact tests. Continuous variables will be evaluated by a two-sample t-test, a 95% confidence interval and p-value will be reported.

   For time-dependent analyses, Hazard Ratios will be evaluated using Cox proportional hazards model and Kaplan Meier estimates will be evaluated according to log-rank test.

   1.4 Missing Data.

   Every effort will be undertaken to minimize missing data. The following approach to handling missing data will be adopted based on the type of the outcome and endpoint being analyzed.

   Kaplan-Meier estimates will censor incomplete data at the last date of available follow-up information, assuming complete reporting of all events up to that date and event status unknown after that date.

   1.5 Calculating Days to Event.

   When calculating the days-to-event, the date the event took place will always be compared to the index procedure date, also in case a staged procedure took place.

   1.6 Within Patient Correlation.

   In case for a patient more than one lesion will be analyzed, in-patient correlation will be taken into account.
2. Study Data Reporting, Monitoring and Quality Assurance.

2.1 Data Recording.

The data collection tool for this study is a validated electronic data capture system that contains a system generated audit trail. Data required according to this protocol are recorded by investigational site personnel via data entry into the internet based Electronic Data Capture (EDC) software system. All internal and external investigational site personnel seeking access must go through a training process before they are granted access to the electric Case Report Form (eCRF). Training records are maintained. All personnel with access to the eCRF are supported by a Service Desk (if applicable).

Clinical data management will be performed in accordance with applicable sponsor's/Clinical Research Organization (CRO)'s standards and data cleaning procedures. This is applicable for data recorded in the eCRF as well as for data from other sources (e.g. laboratory, ECG, adjudication committees).

Edit checks and queries will be built into the EDC application as described in the Data Management Plan. Queries generated by rules and raised by reviewers will be generated and resolved within the EDC application. During this review, subject data will be checked for consistency, omissions, and any apparent discrepancies.

All Adverse Events, medication and medical histories (if applicable) will be coded using Medical Dictionary for Regulatory Activities (MedDRA).

Data received from external sources such as central labs will be reconciled to the clinical database.

Serious Adverse Events in the clinical database will be reconciled with the safety database.

2.2 Source Documentation.

It is the investigator's responsibility that data entries made in the eCRF are supported by source documents maintained for all subjects enrolled in this study.

Source documents include all recordings and observations or notations of clinical activities and all reports and records necessary for the evaluation of the clinical study. The site must implement processes to ensure availability of all required source documentation.

2.3 Monitoring.

Monitoring the clinical investigation at the study site is the responsibility of the monitoring organization through trained and qualified Clinical Research Associates (CRAs). Monitoring will be performed as described in the Monitoring Plan.

2.4 Audit and Inspection.

To ensure compliance with Good Clinical Practices (GCP) and regulatory requirements, a member of the sponsor's (or a designated CRO's) quality assurance unit may arrange to conduct audits to assess the performance of the study at the study sites and of the study documents originating there. The investigator/institution will be informed of the audit outcome.

In addition, inspections by regulatory health authority representatives and Institutional Review Board (IRB) are possible. The investigator should notify the sponsor immediately of any such inspection.

The investigator/institution agrees to allow the auditor or inspector direct access to all relevant documents and allocate his/her time and the time of his/her staff to the auditor/inspector to discuss findings and any issues. Audits and inspections may occur at any time during or after completion of the study.

In accordance with GCP and the Sponsor's audit plans, this study may be selected for audit by representatives from Sponsor. Inspection of site facilities (e.g., pharmacy, Device storage areas, laboratories etc.) and review of study related records will occur in order to evaluate the study conduct and compliance with the protocol, GCP, and applicable regulatory requirements.

2.5 Archiving.

All Case Report Forms (CRFs), study records, reports and source documents that support the CRFs must be retained in the files of the responsible Investigators for a minimum 2 years following notification by the Sponsor or designee that all investigations have been completed, and will further be retained in accordance with local and international guidelines as identified in the clinical study agreement. This documentation must be accessible upon request by international regulatory authorities, the Sponsor (or designee). The sponsor or designee, must approve archiving or transfer of the documentation for relocation purpose of premises, in writing, prior to the actual file transfer. The investigator must notify the Sponsor, in writing, of transfer location, duration, and the procedure for accessing study documentation. The Investigator must contact the Sponsor, or designee, before the destruction of any records and reports pertaining to the study to ensure they no longer need to be retained.

If the Investigator retires, relocates, or for other reasons withdraws from assuming primary responsibility for keeping the study records, custody per written notice must be submitted to the Sponsor, or designee, indicating the name and address of the person accepting primary responsibility. The Ethics Committee (EC) must be notified in writing of the name and address of the new custodian.

2.6 Deviations from Protocol.

A protocol deviation is defined as an event where the study is not conducted according to the protocol and applicable regulations. Protocol deviations that will be collected include, but are not limited to the following:

* Failure to obtain informed consent or failure to obtain informed consent prior to study procedures;
* Enrolling a subject who did not meet inclusion criteria, or met exclusion criteria;
* Not completing protocol-required examinations or evaluations.

A Protocol Deviation eCRF needs to be completed separately for each type of deviation and submitted to the Sponsor and any reviewing Regulatory Body, such as the EC as required.

Protocol deviations are reportable to the Sponsor as soon as possible after their occurrence.

2.6.1 Site Non-Compliance.

If excessive protocol deviations are noted, the Sponsor reserves the right to suspend study enrollment until a sufficient system is in place at the site to reduce further deviations, or to withdraw the site from participation in the study.

2.7 Compliance to Standard Regulations.

The protocol, informed consent form and other study-related documents will be submitted to the EC / IRB. The study will be performed in accordance with the Declaration of Helsinki and GCP.

The trial will only start at a clinical site after written approval of the study has been obtained from the appropriate national EC/IRB.

ELIGIBILITY:
Inclusion Criteria:

-

Clinical Inclusion Criteria:

1. Subject must be male or nonpregnant female ≥18 years of age and ≤75 years of age;
2. Subject has symptomatic coronary artery disease with objective evidence of ischemia or silent ischemia;
3. Subject is eligible for PCI;
4. Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed;
5. Subject is willing to comply with all protocol-required follow-up evaluation.

Angiographic Inclusion Criteria:

1. Subjects have coronary bifurcation lesions requiring PCI with stent implantation according to clinical guidelines and/or the operator's judgement;
2. Visually estimated reference vessel diameter (RVD) of target main vessel ≥2.5 mm and ≤4.0 mm;
3. Visually estimated RVD of target side branch ≥ 2.0mm;
4. Coronary anatomy is likely to allow delivery of a study device to the target lesion(s);
5. V-RESOLVE score ≥ 12 points.

Exclusion Criteria:

-

Clinical Exclusion Criteria:

1. Subject has a known allergy to contrast (that cannot be adequately pre-medicated) and/or the trial stent system or protocol-required concomitant medications (e.g., stent alloy, stainless steel, sirolimus, everolimus or structurally related compounds, polymer or individual components, all P2Y12 inhibitors, or aspirin);
2. Planned surgery within 6 months after the index procedure;
3. Subject has one of the following (as assessed prior to the index procedure):

   * Other serious medical illness (e.g., cancer, congestive heart failure) with estimated life expectancy of less than 12 months；
   * Current problems with substance abuse (e.g., alcohol, cocaine, heroin, etc.);
   * Planned procedure that may cause non-compliance with the protocol or confound data interpretation;
4. Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions;
5. Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint;
6. Subject intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure;
7. Subject with known intention to procreate within 12 months after the index procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure);
8. Subject is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential);
9. Subject with left ventricular ejection fraction < 35%;
10. Subject has preoperative renal dysfunction: serum creatinine>2.0mg/dl (176.82umol/L).

Angiographic Exclusion Criteria:

1. Left main lesions;
2. In case of acute myocardial infarction of which the culprit vessel located at the left anterior descending (LAD) artery, the bifurcation lesion (LAD/diagonal branch [RVD>2.5mm]) which is proximal to occluded LAD segment should be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
side branch occlusion after main vessel stenting | Immediately after the main vessel
  The primary endpoint is side branch occlusion, which is defined as any decrease in TIMI flow grade or absence of flow in side branch after main vessel stent well opposed.

SECONDARY OUTCOMES:
The elevation of biomarkers of peri-procedural myocardial injury (Creatine Kinase-Myocardial Band (CK-MB) and Troponin I) | 48h after Percutaneous Coronary Intervention (PCI)
  Peri-procedural Myocardial Infarction (MI) is defined as biomarkers elevation ≥10 × upper reference limit (URL) for CK-MB and/or ≥70 × URL for troponin.
Major adverse cardiac events (MACE) | 12-month
  Including all cause death, all myocardial infarction (MI) and target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Kefei Dou, MD, PhD, Principal Investigator — Fuwai Hospital and National Center for Cardiovascular Diseases; Bo Xu, MBBS, Principal Investigator — Fuwai Hospital and National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Iakovou I, Schmidt T, Bonizzoni E, Ge L, Sangiorgi GM, Stankovic G, Airoldi F, Chieffo A, Montorfano M, Carlino M, Michev I, Corvaja N, Briguori C, Gerckens U, Grube E, Colombo A. Incidence, predictors, and outcome of thrombosis after successful implantation of drug-eluting stents. JAMA. 2005 May 4;293(17):2126-30. doi: 10.1001/jama.293.17.2126. PMID 15870416
- [Background] Steigen TK, Maeng M, Wiseth R, Erglis A, Kumsars I, Narbute I, Gunnes P, Mannsverk J, Meyerdierks O, Rotevatn S, Niemela M, Kervinen K, Jensen JS, Galloe A, Nikus K, Vikman S, Ravkilde J, James S, Aaroe J, Ylitalo A, Helqvist S, Sjogren I, Thayssen P, Virtanen K, Puhakka M, Airaksinen J, Lassen JF, Thuesen L; Nordic PCI Study Group. Randomized study on simple versus complex stenting of coronary artery bifurcation lesions: the Nordic bifurcation study. Circulation. 2006 Oct 31;114(18):1955-61. doi: 10.1161/CIRCULATIONAHA.106.664920. Epub 2006 Oct 23. PMID 17060387
- [Background] Genereux P, Kumsars I, Lesiak M, Kini A, Fontos G, Slagboom T, Ungi I, Metzger DC, Wykrzykowska JJ, Stella PR, Bartorelli AL, Fearon WF, Lefevre T, Feldman RL, LaSalle L, Francese DP, Onuma Y, Grundeken MJ, Garcia-Garcia HM, Laak LL, Cutlip DE, Kaplan AV, Serruys PW, Leon MB. A randomized trial of a dedicated bifurcation stent versus provisional stenting in the treatment of coronary bifurcation lesions. J Am Coll Cardiol. 2015 Feb 17;65(6):533-43. doi: 10.1016/j.jacc.2014.11.031. PMID 25677311
- [Background] Chen SL, Santoso T, Zhang JJ, Ye F, Xu YW, Fu Q, Kan J, Paiboon C, Zhou Y, Ding SQ, Kwan TW. A randomized clinical study comparing double kissing crush with provisional stenting for treatment of coronary bifurcation lesions: results from the DKCRUSH-II (Double Kissing Crush versus Provisional Stenting Technique for Treatment of Coronary Bifurcation Lesions) trial. J Am Coll Cardiol. 2011 Feb 22;57(8):914-20. doi: 10.1016/j.jacc.2010.10.023. PMID 21329837
- [Background] Abdel-Latif A, Moliterno DJ. Bifurcation stenting techniques and outcomes in patients with stable coronary artery disease: more evidence suggesting simpler is safer. JACC Cardiovasc Interv. 2015 Apr 20;8(4):561-3. doi: 10.1016/j.jcin.2015.02.004. No abstract available. PMID 25907083
- [Background] Hahn JY, Chun WJ, Kim JH, Song YB, Oh JH, Koo BK, Rha SW, Yu CW, Park JS, Jeong JO, Choi SH, Choi JH, Jeong MH, Yoon JH, Jang Y, Tahk SJ, Kim HS, Gwon HC. Predictors and outcomes of side branch occlusion after main vessel stenting in coronary bifurcation lesions: results from the COBIS II Registry (COronary BIfurcation Stenting). J Am Coll Cardiol. 2013 Oct 29;62(18):1654-1659. doi: 10.1016/j.jacc.2013.07.041. Epub 2013 Aug 14. PMID 23954335
- [Background] Kralev S, Poerner TC, Basorth D, Lang S, Wolpert C, Haghi D, Borggrefe M, Haase KK, Suselbeck T. Side branch occlusion after coronary stent implantation in patients presenting with ST-elevation myocardial infarction: clinical impact and angiographic predictors. Am Heart J. 2006 Jan;151(1):153-7. doi: 10.1016/j.ahj.2005.01.034. PMID 16368309
- [Background] Aliabadi D, Tilli FV, Bowers TR, Benzuly KH, Safian RD, Goldstein JA, Grines CL, O'Neill WW. Incidence and angiographic predictors of side branch occlusion following high-pressure intracoronary stenting. Am J Cardiol. 1997 Oct 15;80(8):994-7. doi: 10.1016/s0002-9149(97)00591-2. PMID 9352966
- [Background] Latib A, Colombo A. Bifurcation disease: what do we know, what should we do? JACC Cardiovasc Interv. 2008 Jun;1(3):218-26. doi: 10.1016/j.jcin.2007.12.008. PMID 19463303
- [Background] Colombo A, Ruparelia N. When you ask yourself the question "should I protect the side branch?": the answer is "yes". JACC Cardiovasc Interv. 2015 Jan;8(1 Pt A):47-8. doi: 10.1016/j.jcin.2014.11.007. No abstract available. PMID 25616816
- [Background] Singh J, Patel Y, Depta JP, Mathews SJ, Cyrus T, Zajarias A, Kurz HI, Lasala JM, Bach RG. A modified provisional stenting approach to coronary bifurcation lesions: clinical application of the "jailed-balloon technique". J Interv Cardiol. 2012 Jun;25(3):289-96. doi: 10.1111/j.1540-8183.2011.00716.x. Epub 2012 Feb 26. PMID 22364484
- [Background] Burzotta F, Trani C, Sianos G. Jailed balloon protection: a new technique to avoid acute side-branch occlusion during provisional stenting of bifurcated lesions. Bench test report and first clinical experience. EuroIntervention. 2010 Feb;5(7):809-13. doi: 10.4244/eijv5i7a135. PMID 20142195
- [Background] Muramatsu T, Onuma Y, Garcia-Garcia HM, Farooq V, Bourantas CV, Morel MA, Li X, Veldhof S, Bartorelli A, Whitbourn R, Abizaid A, Serruys PW; ABSORB-EXTEND Investigators. Incidence and short-term clinical outcomes of small side branch occlusion after implantation of an everolimus-eluting bioresorbable vascular scaffold: an interim report of 435 patients in the ABSORB-EXTEND single-arm trial in comparison with an everolimus-eluting metallic stent in the SPIRIT first and II trials. JACC Cardiovasc Interv. 2013 Mar;6(3):247-57. doi: 10.1016/j.jcin.2012.10.013. PMID 23517836
- [Background] Moussa ID, Klein LW, Shah B, Mehran R, Mack MJ, Brilakis ES, Reilly JP, Zoghbi G, Holper E, Stone GW. Consideration of a new definition of clinically relevant myocardial infarction after coronary revascularization: an expert consensus document from the Society for Cardiovascular Angiography and Interventions (SCAI). J Am Coll Cardiol. 2013 Oct 22;62(17):1563-70. doi: 10.1016/j.jacc.2013.08.720. PMID 24135581
- [Result] Dou K, Zhang D, Xu B, Yang Y, Yin D, Qiao S, Wu Y, Yan H, You S, Wang Y, Wu Z, Gao R, Kirtane AJ. An angiographic tool for risk prediction of side branch occlusion in coronary bifurcation intervention: the RESOLVE score system (Risk prEdiction of Side branch OccLusion in coronary bifurcation interVEntion). JACC Cardiovasc Interv. 2015 Jan;8(1 Pt A):39-46. doi: 10.1016/j.jcin.2014.08.011. PMID 25616815
- [Derived] Zhang D, Zhao Z, Gao G, Xu H, Wang H, Liu S, Yin D, Feng L, Zhu C, Wang Y, Zhao Y, Yang Y, Gao R, Xu B, Dou K. Jailed Balloon Technique Is Superior to Jailed Wire Technique in Reducing the Rate of Side Branch Occlusion: Subgroup Analysis of the Conventional Versus Intentional StraTegy in Patients With High Risk PrEdiction of Side Branch OccLusion in Coronary Bifurcation InterVEntion Trial. Front Cardiovasc Med. 2022 Mar 31;9:814873. doi: 10.3389/fcvm.2022.814873. eCollection 2022. PMID 35433861
- [Derived] Dou K, Zhang D, Pan H, Guo N, Li L, Li Y, Zhang Q, Liu B, Shen Z, Zhang B, Liu J, Han W, Wang Y, Zhao Y, Yang Y, Chen S, Xie L, Guan C, Kirtane AJ, Xu B; CIT-RESOLVE Investigators. Active SB-P Versus Conventional Approach to the Protection of High-Risk Side Branches: The CIT-RESOLVE Trial. JACC Cardiovasc Interv. 2020 May 11;13(9):1112-1122. doi: 10.1016/j.jcin.2020.01.233. PMID 32381188
- [Derived] Zhang D, Yin D, Song C, Zhu C, Kirtane AJ, Xu B, Dou K. A randomised comparison of Conventional versus Intentional straTegy in patients with high Risk prEdiction of Side branch OccLusion in coronary bifurcation interVEntion: rationale and design of the CIT-RESOLVE trial. BMJ Open. 2017 Jun 12;7(6):e016044. doi: 10.1136/bmjopen-2017-016044. PMID 28606906